CLINICAL TRIAL: NCT05292079
Title: CAPTURER PMCF Post-Market Clinical Follow-up Study
Brief Title: CAPTURER PMCF Study ( rEPIC04D )
Acronym: rEPIC04D
Status: Completed | Type: Observational
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Other Study IDs: CAPTURER PMCF Study
Record Dates: First submitted 2022-03-14; First posted 2022-03-23 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease (CAD); Ischemic Heart Disease
Keywords: MDR (Medical Device Regulations); PMCF (Post-Market Clinical Follow-up); Thrombus extraction catheter
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Coronary Artery Disease (CAD)
  Interventions: Device: CAPTURER

INTERVENTIONS:
Device: CAPTURER — Patients in whom treatment with (CAPTURER) has been attempted

SUMMARY:
Multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study to confirm and support the clinical safety and performance of CAPTURER to meet EU Medical Device regulation (MDR) requirements in all the CONSECUTIVE patients treated with CAPTURER .

DETAILED DESCRIPTION:
The objective of this multicenter, prospective, non-randomized, post-market clinical follow-up (PMCF) study is to confirm and support the clinical safety and performance of the CAPTURER in a NON-SELECTED, Real World population under daily clinical practice when used as intended by the manufacturer to meet EU Medical Device regulation requirements for post-market clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated with CAPTURER according to routine hospital practice and following instructions for use
* Informed consent signed

Exclusion Criteria:

* Not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated with CAPTURER according to routine hospital practice and following instructions for use
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2022-09-29 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2023-12-27 (Actual)

PRIMARY OUTCOMES:
Safety Endpoint. Freedom from Target Lesion Failure | 30 days
  Freedom from TARGET LESION FAILURE (TLF), composite end point of cardiac death, myocardial infarction, stroke and and new Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
Efficacy Endpoint. Freedom from Target Lesion Failure | 30 days
  Freedom from TARGET LESION FAILURE (TLF), composite endpoint of cardiac death, myocardial infarction (MI) and and new Target Lesion Revascularization (TLR)
Freedom from Device rupture | During percutaneous coronary intervention (PCI)
  Freedom from Device rupture
Freedom from Kinking | During PCI
  Freedom from Kinking
Freedom from Complicated withdrawal | During PCI
  Freedom from Complicated withdrawal
Freedom from Coronary perforation | During PCI
  Freedom from Coronary perforation
Freedom from Coronary dissection >C | During PCI
  Freedom from Coronary dissection >C
Freedom from No reflow | During PCI
  Freedom from No reflow
Freedom from Coronary thrombosis | During PCI
  Freedom from Coronary thrombosis

CONTACTS AND LOCATIONS:
Locations (5):
- Spain (5):
  - H. Puerta Del Mar, Cadiz
  - Hospital de San Pedro, Logroño
  - Hospital Universitario Regional de Malaga, Málaga
  - Hospital Universitario Virgen de La Victoria, Málaga
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela

REFERENCES:
- [Background] Gruntzig A. Transluminal dilatation of coronary-artery stenosis. Lancet. 1978 Feb 4;1(8058):263. doi: 10.1016/s0140-6736(78)90500-7. No abstract available. PMID 74678
- [Background] Chevalier B, Gilard M, Lang I, Commeau P, Roosen J, Hanssen M, Lefevre T, Carrie D, Bartorelli A, Montalescot G, Parikh K. Systematic primary aspiration in acute myocardial percutaneous intervention: a multicentre randomised controlled trial of the export aspiration catheter. EuroIntervention. 2008 Aug;4(2):222-8. doi: 10.4244/eijv4i2a40. PMID 19110787
- [Background] Svilaas T, Vlaar PJ, van der Horst IC, Diercks GF, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Thrombus aspiration during primary percutaneous coronary intervention. N Engl J Med. 2008 Feb 7;358(6):557-67. doi: 10.1056/NEJMoa0706416. PMID 18256391
- [Background] Sardella G, Mancone M, Bucciarelli-Ducci C, Agati L, Scardala R, Carbone I, Francone M, Di Roma A, Benedetti G, Conti G, Fedele F. Thrombus aspiration during primary percutaneous coronary intervention improves myocardial reperfusion and reduces infarct size: the EXPIRA (thrombectomy with export catheter in infarct-related artery during primary percutaneous coronary intervention) prospective, randomized trial. J Am Coll Cardiol. 2009 Jan 27;53(4):309-15. doi: 10.1016/j.jacc.2008.10.017. PMID 19161878